CLINICAL TRIAL: NCT04475835
Title: Study on Safety and Efficacy of Bivalirudin During Short-term Intervention of Non-infarction Related Artery for Acute ST-segment Elevation Myocardial Infarction After Emergency Percutaneous Coronary Intervention
Brief Title: Safety and Efficacy of Bivalirudin During Short-term Intervention of Non-infarction Related Artery After PPCI of STEMI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XJTU1AF2020LSK-017
Record Dates: First submitted 2020-07-15; First posted 2020-07-17 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: STEMI With Multivessel Coronary Disease
MeSH Terms: interventions — bivalirudin; Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bivalirudin (Experimental): Bivalirudin with prolonged full dose infusion during PCI
  Interventions: Drug: Bivalirudin
- Heparin (Active Comparator): Heparin 100U/kg
  Interventions: Drug: Heparin

INTERVENTIONS:
Drug: Bivalirudin — Bivaliruding 0.75 mg/kg intravenous bolus loading dose, and immediately followed by intravenous infusion of 1.75 mg/kg/h until 4 hours after PCI. A prolonged infusion of 0.2 mg/kg/h for ≤20h could be considered at the operator's discretion. It is recommended that ACT be monitored 5 minutes after the first administration, and if ACT is <225 s (Hemotec method), intravenous injection of 0.30 mg/kg of bivalirudin should be administered.
  Arms: Bivalirudin
Drug: Heparin — Heparin is dosed at 100 U/kg. ACT is monitored 5 min after the first administration, and if the ACT <225 s (Hemotec method), an intravenous injection of heparin should be administered by need.
  Arms: Heparin

SUMMARY:
This is a randomized, open label, cohort study, in which a total of 100 patients will be enrolled and randomly assigned to receive bivalirudin or heparin in a 1:1 ratio during short-term intervention of non-infarction related artery for acute ST-segment elevation myocardial infarction after emergency percutaneous coronary intervention.

NACE, MACE, any type of BARC bleeding, stent thrombosis will be evaluated in 30 days and 6 months after recruitment.

DETAILED DESCRIPTION:
The 2017 guideline gives a class IIA recommendation ('should be considered') for complete revascularisation in patients presenting with STEMI and multivessel disease, which is approximately 50% of the STEMI population. Staged multivessel PCI during hospitalization (3-5 days after PPCI) is common in contemporary practice.

Patients undergoing primary PCI should receive enhanced antithrombotic therapy, includes DAPT and and parenteral anticoagulant, which caused an increased bleeding risk. In addition, repeated use of heparin in a short time may increase the incidence of HIT. Direct thrombin inhibitor bivalirudin, demonstrated a reduced risk of bleeding and an overall favorable profile including reduced NACE.

This is a randomized, open label, cohort study, which is aimed to investigate the safety and efficacy of bivalirudin during short-term intervention of non-infarction related artery for acute ST-segment elevation myocardial infarction after emergency percutaneous coronary intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Acute STEMI (including patients within 12 h of symptom onset, or 24-48 h with recurrent or ongoing chest pain chest pain, persistent ST-segment elevation or new left bundle branch block.
* Staged intervention of non-infarction related artery within 5 days after PPCI during Hospitalization.
* Signed informed consent.

Exclusion Criteria:

* Cardiogenic shock.
* Received thrombolytic therapy or used any anticoagulant drugs within 48 hours before randomized.
* Active bleeding, recent bleeding events or bleeding tendency.
* History of surgery in the last 1 month.
* Suspicious symptoms of aortic dissection, pericarditis and endocarditis.
* Blood pressure > 180/110 mmHg.
* Hemoglobin < 100 g/L, Platelet count <100×10(9)/L, Transaminase 3 times upper limit of normality or Creatinine clearance <30ml/min.
* History of Heparin-Induced Thrombocytopenia.
* Allergic to any research drug or device.
* Pregnancy or lactation.
* Any condition that makes the patient unsuitable for PCI or may interfere with the study.
* Patient disagrees or fails to sign the written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-01-12 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Net adverse clinical events (NACE) | 30 days
  A composite of major adverse cardiac or cerebral events (all-cause death, reinfarction, ischemia-driven target vessel revascularization, or stroke) or any bleeding as defined by BARC definition (grades 1-5).
  BARC=Bleeding Academic Research Consortium

SECONDARY OUTCOMES:
Major adverse cardiac and cerebral events (MACE) | 30 days
  A composite of all-cause death, reinfarction, ischemia-driven target vessel revascularization, or stroke
Major adverse cardiac and cerebral events (MACE) | 6 months
  A composite of all-cause death, reinfarction, ischemia-driven target vessel revascularization, or stroke
Bleeding | 30 days
  Bleeding as defined by BARC definition (grades 1-5). Bleeding was considered medically actionable if BARC types 2-5 and was considered major if BARC types 3-5 occurred.
  BARC=Bleeding Academic Research Consortium
Bleeding | 6 months
  Bleeding as defined by BARC definition (grades 1-5). Bleeding was considered medically actionable if BARC types 2-5 and was considered major if BARC types 3-5 occurred.
  BARC=Bleeding Academic Research Consortium
Stent thrombosis | Hospitalization
  Stent thrombosis as defined by ARC ARC=Academic Research Consortium
Stent thrombosis | 30 days
  Stent thrombosis as defined by ARC ARC=Academic Research Consortium
Stent thrombosis | 6 months
  Stent thrombosis as defined by ARC ARC=Academic Research Consortium

CONTACTS AND LOCATIONS:
Overall Officials: Yihui Xiao, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China